CLINICAL TRIAL: NCT03238768
Title: Enhanced Early Nutrition for Preterm Infants to Improve Neurodevelopment and Minimize Metabolic Risk
Brief Title: Enhanced Nutrition for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00000063
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Preterm Birth
Keywords: Nutrition; Body Composition; Preterm; Neonate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Infants will be randomized to receive either standard parenteral nutrition via the NICU protocol or enhanced parenteral nutrition via the Study protocol during their first week of life through higher initial macronutrient provision and faster advancement of macronutrient provision.
Who Masked: Participant, Outcomes Assessor
Masking Description: Parents, participant and Outcomes assessor will be blinded to the nutritional intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Nutrition (Experimental): Infants randomized to the study protocol will start on higher initial amounts of calories, proteins and fats. They will also undergo faster increases of these nutrients during their first week of life.
  Interventions: Other: Enhanced Intravenous Nutrition
- Standard Nutrition (Active Comparator): Infants randomized to the standard nutrition protocol will start on standard amounts of calories, proteins and fats per the usual NICU routine. They will also undergo standard increases of these nutrients during their first week of life.
  Interventions: Other: Standard Intravenous Nutrition

INTERVENTIONS:
Other: Enhanced Intravenous Nutrition — Increased macronutrients for first 7 days
  Arms: Enhanced Nutrition
Other: Standard Intravenous Nutrition — Standard macronutrients for first 7 days
  Arms: Standard Nutrition

SUMMARY:
The overall objective of the proposal is to demonstrate the feasibility of providing increased calories and protein in the first week of life to very low birth weight (VLBW) preterm infants.

DETAILED DESCRIPTION:
Infants will be randomized to receive either standard parenteral nutrition via the neonatal intensive care unit (NICU) protocol or enhanced parenteral nutrition via the Study protocol during their first week of life through higher initial macronutrient provision and faster advancement of macronutrient provision.

ELIGIBILITY:
Inclusion Criteria:

* VLBW (birth weight <1500grams) preterm (gestational age (GA) at birth < 32 weeks) infants admitted to the University of Minnesota Masonic Children's Hospital NICU, for which written informed consent can be secured from a parent within 12 hours of birth.

Exclusion Criteria:

* Infants who are diagnosed prenatally with a clinical condition (other than prematurity) that is known to affect growth rate, adiposity, or neurocognitive development, who experienced severe birth asphyxia, who are enrolled in another study affecting nutritional management, or who are likely to be transferred out of the NICU will be excluded from participation.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the amount of nutrition ( kcals/kg/day and amount of protein g/kg/day and amount of lipids g/kg/day) received in the first week of life. | 1 week
  We will calculate the actual amount of protein, kcals, lipids etc received in both groups at the end of the first week to determine if we were able to deliver increased amounts of nutrition to the enhanced protocol group

CONTACTS AND LOCATIONS:
Overall Officials: Sara E Ramel, MD, Principal Investigator — University of Minnesota Masonic Children's Hospital
Locations (1):
- University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagel EM, Gonzalez V JD, Bye JK, Super J, Demerath EW, Ramel SE. Enhanced Parenteral Nutrition Is Feasible and Safe in Very Low Birth Weight Preterm Infants: A Randomized Trial. Neonatology. 2023;120(2):242-249. doi: 10.1159/000527552. Epub 2023 Feb 22. PMID 36812894

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT03238768/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03238768/ICF_001.pdf